CLINICAL TRIAL: NCT04897997
Title: Effect of Smoking on Activated Clotting Time Values During Coronary Angioplasty
Brief Title: Effect of Smoking on Activated Clotting Time Values During Coronarography and Angioplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Camenzind, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 20210502VandoeuvreFranceEurope
Record Dates: First submitted 2021-05-04; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Ischemic Cardiomyopathy
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sampling
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- non smokers: never having smoked patients
  Interventions: Procedure: coronarography and angioplasty
- smokers: actively smoking patients
  Interventions: Procedure: coronarography and angioplasty
- acute coronary syndrome: patients with the coronary indication of ACS
  Interventions: Procedure: coronarography and angioplasty
- stable: patients with the coronary indication of stable or silent ischemia
  Interventions: Procedure: coronarography and angioplasty

INTERVENTIONS:
Procedure: coronarography and angioplasty — selective angiography of the coronaries and angioplasty of significant culprit lesion(s)

SUMMARY:
analyzing influence of smoking on patients anti-coagulation status as assessed by ACT measurements during coronary angioplasty

DETAILED DESCRIPTION:
During angioplasty, activated clotting time (ACT) measurements are recommended to attest the correct anticoagulation level and if anticoagulation levels are suboptimal after the two first boluses, additional unfractionated heparin (UFH) injections are recommended until obtention of a therapeutic ACT values (250-350s).

The study hypothesis was that the procoagulant effect of the tobacco may be responsible of reduced anticoagulation levels after standardized UFH administrations and thus presenting an UFH resistance requiring increased UFH dosages to obtain a therapeutic ACT values.

ELIGIBILITY:
Inclusion Criteria:

* any patient older than 18 years needing a diagnostic coronarography was eligible for enrollment

Exclusion Criteria:

* unconscious patient
* any patient presenting with one of the following characteristic known to impact either on ACT or aPTT measurements as: oral anticoagulation medication (anti-vitamin K and non-vitamin K antagonist oral anticoagulants [NOAC]), fondaparinux or LMWH usage, coagulopathy defined as prothrombin time < 50 % or thrombopenia < 50 000 G/L, declared or observed thrombophilia defined as antithrombin < 50%, baseline aPTT values with a ratio patient/control > 1.2 presence of lupus anticoagulant, connective tissue disease, active cancer
* a person as defined by the law articles L. 1121-5, L. 1121-7 et L1121-8 of the Code de la santé publique, France (pregnant, parturient women or breastfeeding women, legally adult patient under legal protection measure [tutelage, protection of vulnerable adults]),
* a person as defined by the law articles L. 3212-1 et L. 3213-1 of the Code de la santé publique, France (legally adult patient unable to consent, person with legal or administrative freedom restriction or person under psychiatric treatment)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: any patient needing a coronarography followed by an angioplasty without the above mentioned exclusion criteria
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
ACT values after injection the first injection of a standardized unfractionated heparin bolus between non-smoking and actively smoking patients | during the intervention
  comparison of ACT values after injection of two standardized UFH boluses between non-smoking and actively smoking patients (non-smoker group versus active smoker group)
ACT values after injection the second injection of a standardized unfractionated heparin bolus between non-smoking and actively smoking patients | immediately after the intervention
  comparison of ACT values after injection of two standardized UFH boluses between non-smoking and actively smoking patients (non-smoker group versus active smoker group)

SECONDARY OUTCOMES:
ACT values after injection of the first standardized UFH bolus in ex-smokers | during the intervention
  ACT values after injection of the first standardized UFH bolus in ex-smokers requiring a coronarography followed by a PTCA
ACT values after injection of the second standardized UFH bolus in ex-smokers | immediately after the intervention
  ACT values after injection of the second standardized UFH bolus in ex-smokers requiring a coronarography followed by a PTCA

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Camenzind, Professor, Study Director — University Hospital Nancy France
Locations (1):
- University Hospital Nancy Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No